CLINICAL TRIAL: NCT05299489
Title: Clinical Randomized Controlled Trial To Compare Direct and Indirect Composite Restoration in Children With Molar Incisor Hypomineralization Patients (MIH)
Brief Title: Evaluation Direct and Indirect Composite Restoration in Hypomineralization Molars.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: UDDS-Pedo-10-2022
Record Dates: First submitted 2022-03-04; First posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Dental Enamel Hypoplasia; Dental Caries
Keywords: MIH; Direct composite; Indirect composite; Permanent molars
MeSH Terms: conditions — Dental Enamel Hypoplasia; Dental Caries

STUDY DESIGN:
Intervention Model Description: Split mouth design
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Direct composite in hypomineraliztion molars. (Experimental)
  Interventions: Other: Direct restoration
- Indirect composite in hypomineraliztion molars. (Other)
  Interventions: Other: Indirect restoration

INTERVENTIONS:
Other: Direct restoration — Local anesthesia was achieved and the tooth were isolated using a rubber dam. Then, the entire caries and hypomineralized enamel were removed using diamond burs and removal the affected dentine caries by slow speed handpiece, the final preparation must be on intact enamel. The molars were wiped using 5.25% sodium hypochlorite followed by rinsing with water, etching using 37% phosphoric acid The surface of the restoration, bonding, applying composite and assessment of occlusion.
  Arms: Direct composite in hypomineraliztion molars.
Other: Indirect restoration — Local anesthesia was achieved and the tooth were isolated using a rubber dam. Then, the entire caries and hypomineralized enamel were removed using diamond burs and removal the affected dentine caries by slow speed handpiece, the final preparation must be on intact enamel. Preparation walls were vertical according to the longitudinal axis of the tooth and the occlusal depth 2 mm. The impressions were taken for both jaws and the bite were recorded for the using red wax. The cavity in example were painted with insulating material. Indirect composite resin were applied, finishined and polished.
  Cementation:
  Tooth surface: The molars were wiped using 5.25% sodium hypochlorite followed by rinsing with water, etching using 37% phosphoric acid The surface of the restoration: application of silane coupling agent to enhance the formation of resin tags.
  Dual cure resin cement was used for final cementation followed by an assessment of occlusion.
  Arms: Indirect composite in hypomineraliztion molars.

SUMMARY:
The aim of this study is to evaluate the effectiveness of direct and Indirect Composite Restoration in Children With Molar Incisor Hypomineralization Patients (MIH) and following up after 3 , 6 , 12 months (Clinically):

Group A ( Control group ): Hypomineralization molars were restored by direct composite.

Group B ( Experimental group ): Hypomineralization molars were restored by indirect composite.

DETAILED DESCRIPTION:
Pediatric dentists face a high prevalence of MIH ranging from 3 to 40%, so it is relatively common condition that would cause treatment challenges due to severe sensitivity, breakdown of the occlusal surface, difficulty anesthesia and relatively high failure of restorations as a result of marginal breakdown of restorations.

There are many treatment options available to restore these teeth. In mild and moderate cases, they are restored using direct composite resin. In cases where teeth are severely affected, the treatment is more complicated, including stainless steel crowns and different types of full or partial indirect crowns.

Direct composite resin restorations are the treatment option in the majority of clinical cases, but in severe cases, the results of treatment are often unsatisfactory.

Indirect composite restorations are an aesthetic alternative to cast metal inlays and stainless steel crowns with minimal microleakage.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 8 and 12 years.
2. Definitely positive or positive ratings of Frank scale.
3. The first permanent molars must achieve the following criteria: The molar must be suffering from severe demineralization and it must be restorable with composite.
4. caries lesions include the occlusal surface and should not extend more than thirds of the thickness of dentin
5. Absence clinical and radiographic signs which indicate pulp necrosis

Exclusion Criteria:

1. Systematic or mental disorders.
2. Definitely negative or negative ratings of Frankel scale
3. Existence periapical translucence
4. Existence external or internal abnormal absorption
5. Existence swelling or fistula
6. Sensitivity to percussion
7. Existence of spontaneous or stimulant pain

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-12-25 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Clinical evaluation of teeth restored by direct composite. | 3 months after applying the restoration
  Clinical evaluation of restored tooth was assessed according to USPHS criteria (Alpha, Bravo, Charlie) as following:
  Marginal Adaptation: (No crevice), (Crevice), (Fractured, missing). Marginal Discoloration: (no discoloration), (discoloration but has not penetrated along the margin), (discoloration has present along the). Secondary caries: (No evidence of caries), (Evidence of caries). Color Matching: (100% color match), (Slight mismatched), (Total mismatched). Anatomic Form: (anatomic form), (teeth partially degraded but clinically acceptable), (partially degraded but need to be replaced). Postoperative Sensitivity: (no Postoperative sensitivity), (slight sensitivity), (sever sensitivity).Retention: (no loss) (fracture or loss). Surface Texture: (no defect), (minimal defect), (severed defect).
Clinical evaluation of teeth restored by direct composite. | 6 months after applying the restoration
  Clinical evaluation of restored tooth was assessed according to USPHS criteria (Alpha, Bravo, Charlie) as following:
  Marginal Adaptation: (No crevice), (Crevice), (Fractured, missing). Marginal Discoloration: (no discoloration), (discoloration but has not penetrated along the margin), (discoloration has present along the). Secondary caries: (No evidence of caries), (Evidence of caries). Color Matching: (100% color match), (Slight mismatched), (Total mismatched). Anatomic Form: (anatomic form), (teeth partially degraded but clinically acceptable), (partially degraded but need to be replaced). Postoperative Sensitivity: (no Postoperative sensitivity), (slight sensitivity), (sever sensitivity).Retention: (no loss) (fracture or loss). Surface Texture: (no defect), (minimal defect), (severed defect).
Clinical evaluation of teeth restored by direct composite. | 12 months after applying the restoration
  Clinical evaluation of restored tooth was assessed according to USPHS criteria (Alpha, Bravo, Charlie) as following:
  Marginal Adaptation: (No crevice), (Crevice), (Fractured, missing). Marginal Discoloration: (no discoloration), (discoloration but has not penetrated along the margin), (discoloration has present along the). Secondary caries: (No evidence of caries), (Evidence of caries). Color Matching: (100% color match), (Slight mismatched), (Total mismatched). Anatomic Form: (anatomic form), (teeth partially degraded but clinically acceptable), (partially degraded but need to be replaced). Postoperative Sensitivity: (no Postoperative sensitivity), (slight sensitivity), (sever sensitivity).Retention: (no loss) (fracture or loss). Surface Texture: (no defect), (minimal defect), (severed defect).
Clinical evaluation of teeth restored by indirect composite. | 3 months after applying the restoration
  Clinical evaluation of restored tooth was assessed according to USPHS criteria (Alpha, Bravo, Charlie) as following:
  Marginal Adaptation: (No crevice), (Crevice), (Fractured, missing). Marginal Discoloration: (no discoloration), (discoloration but has not penetrated along the margin), (discoloration has present along the). Secondary caries: (No evidence of caries), (Evidence of caries). Color Matching: (100% color match), (Slight mismatched), (Total mismatched). Anatomic Form: (anatomic form), (teeth partially degraded but clinically acceptable), (partially degraded but need to be replaced). Postoperative Sensitivity: (no Postoperative sensitivity), (slight sensitivity), (sever sensitivity).Retention: (no loss) (fracture or loss). Surface Texture: (no defect), (minimal defect), (severed defect).
Clinical evaluation of teeth restored by indirect composite. | 6 months after applying the restoration
  Clinical evaluation of restored tooth was assessed according to USPHS criteria (Alpha, Bravo, Charlie) as following:
  Marginal Adaptation: (No crevice), (Crevice), (Fractured, missing). Marginal Discoloration: (no discoloration), (discoloration but has not penetrated along the margin), (discoloration has present along the). Secondary caries: (No evidence of caries), (Evidence of caries). Color Matching: (100% color match), (Slight mismatched), (Total mismatched). Anatomic Form: (anatomic form), (teeth partially degraded but clinically acceptable), (partially degraded but need to be replaced). Postoperative Sensitivity: (no Postoperative sensitivity), (slight sensitivity), (sever sensitivity).Retention: (no loss) (fracture or loss). Surface Texture: (no defect), (minimal defect), (severed defect).
Clinical evaluation of teeth restored by indirect composite. | 12 months after applying the restoration
  Clinical evaluation of restored tooth was assessed according to USPHS criteria (Alpha, Bravo, Charlie) as following:
  Marginal Adaptation: (No crevice), (Crevice), (Fractured, missing). Marginal Discoloration: (no discoloration), (discoloration but has not penetrated along the margin), (discoloration has present along the). Secondary caries: (No evidence of caries), (Evidence of caries). Color Matching: (100% color match), (Slight mismatched), (Total mismatched). Anatomic Form: (anatomic form), (teeth partially degraded but clinically acceptable), (partially degraded but need to be replaced). Postoperative Sensitivity: (no Postoperative sensitivity), (slight sensitivity), (sever sensitivity).Retention: (no loss) (fracture or loss). Surface Texture: (no defect), (minimal defect), (severed defect).

CONTACTS AND LOCATIONS:
Overall Officials: Abdulrhman S Hakmi, Principal Investigator — MSc student in Pedodontics, University of Damascus; Mayssoon Dashash, Phd, Study Director — Professor of Pedodontics, Department of Pedodontics, University of Damascus
Locations (1):
- Damascus University, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weerheijm KL. Molar incisor hypomineralization (MIH): clinical presentation, aetiology and management. Dent Update. 2004 Jan-Feb;31(1):9-12. doi: 10.12968/denu.2004.31.1.9. PMID 15000003
- [Background] Silva MJ, Scurrah KJ, Craig JM, Manton DJ, Kilpatrick N. Etiology of molar incisor hypomineralization - A systematic review. Community Dent Oral Epidemiol. 2016 Aug;44(4):342-53. doi: 10.1111/cdoe.12229. Epub 2016 Apr 28. PMID 27121068
- [Background] Melin L, Lundgren J, Malmberg P, Noren JG, Taube F, Cornell DH. XRMA and ToF-SIMS Analysis of Normal and Hypomineralized Enamel. Microsc Microanal. 2015 Apr;21(2):407-21. doi: 10.1017/S1431927615000033. Epub 2015 Feb 12. PMID 25674916
- [Background] Lygidakis NA, Wong F, Jalevik B, Vierrou AM, Alaluusua S, Espelid I. Best Clinical Practice Guidance for clinicians dealing with children presenting with Molar-Incisor-Hypomineralisation (MIH): An EAPD Policy Document. Eur Arch Paediatr Dent. 2010 Apr;11(2):75-81. doi: 10.1007/BF03262716. PMID 20403301
- [Background] Dhareula A, Goyal A, Gauba K, Bhatia SK, Kapur A, Bhandari S. A clinical and radiographic investigation comparing the efficacy of cast metal and indirect resin onlays in rehabilitation of permanent first molars affected with severe molar incisor hypomineralisation (MIH): a 36-month randomised controlled clinical trial. Eur Arch Paediatr Dent. 2019 Oct;20(5):489-500. doi: 10.1007/s40368-019-00430-y. Epub 2019 Mar 19. PMID 30888581
- [Background] Gaton-Hernandez P, Serrano CR, da Silva LAB, de Castaneda ER, da Silva RAB, Pucinelli CM, Manton D, Ustrell-Torrent JM, Nelson-Filho P. Minimally interventive restorative care of teeth with molar incisor hypomineralization and open apex-A 24-month longitudinal study. Int J Paediatr Dent. 2020 Jan;30(1):4-10. doi: 10.1111/ipd.12581. Epub 2019 Oct 24. PMID 31593607